CLINICAL TRIAL: NCT07269704
Title: Effect of Nutritional Supplement Alpha-ketoglutarate for Age-related Ocular Disease: An Open Label, Single Arm Study to Evaluate the Effect of Alpha-ketoglutarate Administered Orally in Patients With Age-related Ocular Diseases (Metabolic Eye Therapy)
Brief Title: Effect of Nutritional Supplement Alpha-ketoglutarate for Age-related Ocular Disease
Acronym: OAK AGE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Vinit Mahajan, Professor of Ophthalmology, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 68157
Record Dates: First submitted 2025-11-25; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-10

CONDITIONS: Eye Diseases
MeSH Terms: conditions — Eye Diseases | interventions — Ketoglutaric Acids

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Calcium alpha-ketoglutarate (Ca-aKG) (Experimental): At the first and second cataract surgery of the participant, a small amount of tissue (eye fluid ~0.1 ml or 1-2 drops) is removed for analysis. Beginning one week (7 days) prior to their second cataract extraction surgery, the patient takes an oral nutritional supplement (calcium alpha-ketoglutarate) 2 times a day.
  Interventions: Drug: Calcium alpha-ketoglutarate

INTERVENTIONS:
Drug: Calcium alpha-ketoglutarate — Participants took 2 g/day of calcium alpha-ketoglutarate orally, twice daily, for 7 days.
  Other Names: Prohealth Longevity

SUMMARY:
The aims of the study are as follows:

1. Determine how the eye absorbs supplements taken orally.
2. Look for specific signs in the proteins and substances in the eyes of people with eye diseases who are also taking nutritional supplements.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to give written informed consent
2. Able to attend all study visits and complete the study procedures
3. Women of child-bearing potential must have a negative pregnancy test within 2 weeks before cataract surgery. A pregnancy test is not required for postmenopausal women (defined as being at least 12 consecutive months without menses) or those surgically sterilized (those having a bilateral tubal ligation/bilateral salpingectomy, bilateral tubal occlusive procedure, hysterectomy, or bilateral oophorectomy).

Exclusion Criteria:

1. Diabetes and/or thyroid, liver, kidney, bowel, and metabolic diseases or disorders
2. History of supplement allergy or planned major surgery
3. Received any other clinical trial drug within 4 months
4. Calculated creatinine clearance of less than 30 ml/min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2023-08-15 (Actual); Primary Completion 2025-06-10 (Actual); Study Completion 2025-06-10 (Actual)

PRIMARY OUTCOMES:
Mean change in aqueous humor aKG concentration | Baseline and post-supplementation, approximately 28 days
  To evaluate the mean difference in fold-change in aKG levels from baseline to post-supplementation in eye fluid

SECONDARY OUTCOMES:
Mean fold-change in metabolic and retinal pathways | Baseline and post-supplementation, approximately 28 days
  To calculate mean fold-change in retinal metabolic and protein pathways from baseline to post-supplementation in eye fluid

CONTACTS AND LOCATIONS:
Overall Officials: Vinit Mahajan, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Byers Eye Institute, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Age, sex, BMI, Medical history, ocular history
Supporting Information: Study Protocol, ICF
Time Frame: The data will be made available upon study registration with CTgov, and will remain available for at least 5 years.
Access Criteria: Results

REFERENCES:
- [Background] Filip RS, Pierzynowski SG, Lindegard B, Wernerman J, Haratym-Maj A, Podgurniak M. Alpha-ketoglutarate decreases serum levels of C-terminal cross-linking telopeptide of type I collagen (CTX) in postmenopausal women with osteopenia: six-month study. Int J Vitam Nutr Res. 2007 Mar;77(2):89-97. doi: 10.1024/0300-9831.77.2.89. PMID 17896582
- [Background] Riedel E, Nundel M, Hampl H. alpha-Ketoglutarate application in hemodialysis patients improves amino acid metabolism. Nephron. 1996;74(2):261-5. doi: 10.1159/000189319. PMID 8893139
- [Background] Wert KJ, Velez G, Kanchustambham VL, Shankar V, Evans LP, Sengillo JD, Zare RN, Bassuk AG, Tsang SH, Mahajan VB. Metabolite therapy guided by liquid biopsy proteomics delays retinal neurodegeneration. EBioMedicine. 2020 Feb;52:102636. doi: 10.1016/j.ebiom.2020.102636. Epub 2020 Feb 3. PMID 32028070
- [Background] Hou XW, Wang Y, Pan CW. Metabolomics in Age-Related Macular Degeneration: A Systematic Review. Invest Ophthalmol Vis Sci. 2020 Dec 1;61(14):13. doi: 10.1167/iovs.61.14.13. PMID 33315052